CLINICAL TRIAL: NCT01893814
Title: Benefit and Tolerability of a Probiotic Product in Infants With Abdominal Discomfort
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: Probi AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PAB/029911
Record Dates: First submitted 2013-07-02; First posted 2013-07-09 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Abdominal Discomfort
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotics (Active Comparator)
  Interventions: Dietary Supplement: Probiotics
- Control (Placebo Comparator)
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Probiotics
  Arms: Probiotics
Dietary Supplement: Control
  Arms: Control

SUMMARY:
To demonstrate benefit and tolerability of a probiotic product in infants with abdominal discomfort.

ELIGIBILITY:
Inclusion Criteria:

* Male or female singleton
* ≥ 2 weeks and ≤ 12 weeks of age
* Exclusively breastfed at screening
* Abdominal discomfort (infant colic) in the week prior to enrollment, according to the statement of the parent(s) and/or guardian(s)
* Episodes of fussy crying that lasted at least 3 hours a day for at least 3 days in the 7 days prior to enrollment, according to the statement of the parent(s) and/or guardian(s)
* Voluntary, written informed consent of the parent(s) and/or guardian(s) to participate in the study
* Born at full term (37-42 after last menstruation period)
* Birth weight: 2500 - 4500 g
* Weight-for-age ≥ 3th and ≤ 97th percentile according to WHO growth tables / charts
* Apparently healthy at birth (Apgar ≥ 8) and at screening visit
* No major complications during pregnancy or at birth
* Mother 19-45 years of age at childbirth
* Ability of parent(s) and/or guardian(s) to attend visits, interviews and willingness to fill out questionnaires

Exclusion Criteria:

* Intolerance to investigational product/its ingredients
* Severe medical condition or illness, congenital abnormality
* Gastrointestinal disorders (e.g. reflux esophagitis)
* Intake of probiotics and/or antibiotics in the week preceding recruitment and during the study
* Formula feeding at screening/randomisation
* Allergy or atopic disease (family history)
* Participation in another study
* Mother's health condition that may interfere with her ability to take care of her infant
* Mother affected by hepatitis B, HIV or Guillain-Barré Syndrome
* Use of antibiotics by the mother in the week

Ages: 2 Weeks to 12 Weeks | Sex: All
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2013-04; Primary Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Reduction of abdominal discomfort as assessed by comparison of crying time | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Charité Virchow Hospital, Berlin, Germany